CLINICAL TRIAL: NCT04923334
Title: Nonpharmacologic Pain Management in FQHC Primary Care Clinics
Acronym: BeatPain Utah
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Duke University (Other)
Responsible Party: Principal Investigator, Julie Fritz, Distinguished Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00143493
Record Dates: First submitted 2021-06-01; First posted 2021-06-11 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Low Back Pain; Chronic Pain
Keywords: Telehealth; Pain Management; Physical Therapy; Health Disparities
MeSH Terms: conditions — Low Back Pain; Chronic Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: The study design is a clinical trial testing adaptive interventions. All participants receive the Brief Pain Teleconsult in Phase I. We will randomly assign participants with 1:1 distribution to also receive 10-week Telehealth Physical Therapy during Phase I. All participants are re-assessed at 12 weeks and responder status is determined. For participants not receiving Telehealth Physical Therapy in Phase I, further treatment is based on responder status. Responders receive no further treatment. Non-responders receive the 10-week Telehealth Physical Therapy in Phase II. Participants randomized to Telehealth PT in Phase I receive no further treatment. Long-term assessments occur 26 and 52 weeks after randomization.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The study is outcome assessor and investigator blinded. Blinding will only be broken in emergency situations for reasons of participant safety such as a serious adverse event. If blinding is broken, either intentionally or unintentionally, the reason will be fully documented and entered on an electronic case report form. Every effort will be made to discuss the decision to break blinding with the Data Safety Monitoring Board in advance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Pain Teleconsult (Experimental): Participants randomized to Brief Pain Teleconsult will receive the brief teleconsult intervention in Phase 1 (1-12 weeks) Responder status to the Phase 1 treatment will be examined at the 12 week assessment. Participants determined to be non-responders will receive the Telehealth Physical Therapy intervention. Responders receive no additional treatment.
  Interventions: Behavioral: Brief Pain Teleconsult; Behavioral: Telehealth Physical Therapy
- Brief Pain Teleconsult plus Telehealth Physical Therapy (Experimental): Participants randomized to Brief Pain Teleconsult plus Telehealth Physical Therapy will receive the brief teleconsult intervention in Phase 1 followed by the 10-week physical therapy intervention. No additional treatment is provided after the 12 week assessment.
  Interventions: Behavioral: Brief Pain Teleconsult; Behavioral: Telehealth Physical Therapy

INTERVENTIONS:
Behavioral: Brief Pain Teleconsult — The Brief Pain Teleconsult intervention includes 2 sessions provided by a licensed physical therapist over about 1 week. The sessions focus on pain education from a biopsychosocial perspective that is designed to address negative pain appraisals and catastrophizing thoughts, providing advice to be active and engage in exercise and physical activity, and reassurance that activity is beneficial and safe.
Behavioral: Telehealth Physical Therapy — The Telehealth Physical Therapy intervention involves weekly telehealth sessions provided over 10 weeks. Telehealth Physical Therapy is provided by a licensed physical therapist. Key components of the intervention include reinforcing biopsychosocial education messages and developing an exercise and physical activity program using cognitive behavioral principles such as goal setting and positive reinforcement. Pain coping strategies including mindful breathing and progressive relaxation techniques will be included.

SUMMARY:
The goal of this study is to improve pain management and reduce opioid reliance for patients with chronic back pain in Utah Federally-Qualified Health Centers (FQHCs). The study compares the effectiveness of nonpharmacologic pain treatments using telehealth to overcome access barriers. We will use automated EHR reminders for electronic referral to teleconsult services. Our project tests adaptive treatments and uses a hybrid type I design - focused on effectiveness outcomes while gathering implementation data to inform future efforts to scale effective strategies.

DETAILED DESCRIPTION:
This randomized clinical trial compares the effectiveness of different strategies to provide efficacious nonpharmacologic interventions to patients with back pain seeking care in FQHCs throughout the state of Utah. The strategies evaluated are designed to overcome the barriers specific to rural and low income communities served by FQHC clinics through innovative use of telehealth resources. The randomized trial will randomize individual participants to one of two interventions strategies, one providing both a brief pain teleconsult with a 10-week telehealth physical therapy, the other uses an adaptive strategy - providing the brief pain teleconsult first, followed by the 10-week telehealth physical therapy only among those non-responsive to the brief teleconsult treatment. We will also evaluate outcomes related to the efforts to implement strategies in FQHC clinics in order to provide valuable information for future efforts to scale effective strategies into other low resource health care settings. Assessments will occur at baseline and after 12-, 26- and 52-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate in English or Spanish
* Age between 18-80
* Visit with an FQHC provider (in-person or via telehealth) in past 90 days
* Back pain has been an ongoing problem for at least the past 3 months, and has been a problem on at least half the days in the past 6 months
* Access to resources necessary to receive telehealth sessions (phone or 2-way video)

Exclusion Criteria:

* Currently pregnant
* Currently involved in active substance use disorder treatment (other than peer support groups, AA, etc.)
* History of spine surgery in past 6 months
* Has a condition restricting participation in physical activity (i.e., unable to ambulate independently (with or without assistive device) for at least 5 minutes.
* Reason for back pain is a fracture or non-musculoskeletal condition (i.e., spinal tumor, inflammatory disorder, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-11-04 (Actual); Primary Completion 2026-06-21 (Estimated); Study Completion 2026-06-21 (Estimated)

PRIMARY OUTCOMES:
PEG-3 | 12 weeks
  The PEG-3 measure includes 3 items evaluating 1) pain severity, and interference of pain with 2) enjoyment and 3) general activity. Item response options range from 0-10. The PEG-3 score is expressed as the mean of all item scores with higher scores indicating greater pain impact

SECONDARY OUTCOMES:
Physical Function | baseline, 12-, 26- and 52-weeks
  The PROMIS short form 6b for physical function uses fixed items from the PROMIS physical function item bank to provide a T-score with population mean = 50 (sd=10).
Sleep Disturbance | baseline, 12-, 26- and 52-weeks
  The PROMIS short form 6a for sleep disturbance uses fixed items from the PROMIS sleep disturbance item bank to provide a T-score with population mean = 50 (sd=10).
Pain Catastrophizing | baseline, 12-, 26- and 52-weeks
  The PSC-6 is a short-form questionnaire evaluating an individual's negative cognitive-affective response to anticipated or actual pain
Pain Self-Efficacy | baseline, 12-, 26- and 52-weeks
  The PSEQ-4 is a short form questionnaire evaluating an individual's confidence in performing activities despite pain
Global Impression of Change | baseline, 12-, 26- and 52-weeks
  The single-item PGIC assesses participants' of change following treatment based on the question: "Since my treatment, my pain is…" with Likert scale response options ranging from (0) "very much worse" to (6) "very much improved".
opioid use | across 52 week follow-up
  Prescription opioid use across the 52-week follow-up will be examined from EHR noting number of prescriptions and days of use.
PEG-3 | baseline, 26- and 52-weeks
  The PEG-3 measure includes 3 items evaluating 1) pain severity, and interference of pain with 2) enjoyment and 3) general activity. Item response options range from 0-10. The PEG-3 score is expressed as the mean of all item scores with higher scores indicating greater pain impact

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Association of Utah Community Health, Salt Lake City, Utah
  - The University of Utah Healthcare System, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared through the HEAL initiative at NIH
Supporting Information: Study Protocol, SAP
Time Frame: Following completion of the data collection

REFERENCES:
- [Background] Fritz JM, Del Fiol G, Gibson B, Wetter DW, Solis V, Bennett E, Thackeray A, Goode A, Lundberg K, Romero A, Ford I, Stevens L, Siaperas T, Morales J, Yack M, Greene T. BeatPain Utah: study protocol for a pragmatic randomised trial examining telehealth strategies to provide non-pharmacologic pain care for persons with chronic low back pain receiving care in federally qualified health centers. BMJ Open. 2022 Nov 9;12(11):e067732. doi: 10.1136/bmjopen-2022-067732. PMID 36351735
- [Background] Fritz JM, Gibson B, Wetter DW, Del Fiol G, Solis V, Ford I, Lundberg K, Thackeray A. Use of implementation mapping in the planning of a hybrid type 1 pragmatic clinical trial: the BeatPain Utah study. Implement Sci Commun. 2024 Jan 5;5(1):3. doi: 10.1186/s43058-023-00542-z. PMID 38183154
- [Background] Fritz JM, Ford I, George SZ, Vinci de Vanegas L, Cope T, Burke CA, Goode AP. Telehealth delivery of physical therapist-led interventions for persons with chronic low back pain in underserved communities: lessons from pragmatic clinical trials. Front Pain Res (Lausanne). 2024 Apr 19;5:1324096. doi: 10.3389/fpain.2024.1324096. eCollection 2024. PMID 38706872
- [Derived] Fritz JM, Gibson B, Wetter DW, Fiol GD, Solis VH, Ford I, Lundberg K, Thackeray A. Use of implementation mapping in the planning of a hybrid type 1 pragmatic clinical trial: the BeatPain Utah study. Res Sq [Preprint]. 2023 Sep 11:rs.3.rs-3267087. doi: 10.21203/rs.3.rs-3267087/v1. PMID 37790359